CLINICAL TRIAL: NCT03928990
Title: Assesment of Physical Activity Level of Patients With Multiple Sclerosis: From Laboratory to Real Life
Acronym: ACTISEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2018/376
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Device: ActiGraph accelerometer

INTERVENTIONS:
Device: ActiGraph accelerometer — ActiGraph accelerometer + calibration with Cortex MetaMax3B ergospirometer

SUMMARY:
This study aims to assess the feasibility of a protocol determining individual moderate-to-vigorous physical activity (MVPA) thresholds, among multiple sclerosis patients, in routine medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years old
* Multiple sclerosis according to McDonald criteria ;
* Expanded Disability Status Scale (EDSS) between 0 and 6.5 ;
* Patient able to move with or without mechanical assistance.

Exclusion Criteria:

* Deterioration of neurological symptomatology within 60 day before enrollment ;
* Changes brought to the multiple sclerosis treatment within 6 months before enrollment ;
* Introduction of a treatment acting on spasticity or fatigue within 30 day before enrollment
* Changes brought to reeducation protocol throughout the duration of the study
* Patient unable to provide an effort equivalent to 3 times the resting metabolic value = 3 Metabolic Equivalent of Task (METs).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Patient's feeling | Day 1
  Patient's feeling measured at each step of the procedure, measured with Visual Analogique Scale (scored from 0 = not painful to 10 = extremely painful)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France